CLINICAL TRIAL: NCT07120152
Title: A Pharmacokinetic-pharmacodynamic Modeling and Simulation Study of Subcutaneous Infliximab in Patients With Inflammatory Bowel Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Erwin Dreesen (Other)
Collaborators: San Raffaele University Hospital, Italy (Other); University of Liverpool (Other); Hospital Universitario La Fe (Other); University of Southampton (Other); Samsung Medical Center (Other)
Responsible Party: Sponsor-Investigator, Erwin Dreesen, Assistant Professor, KU Leuven
Organization: KU Leuven (Other)
Other Study IDs: G-2024-8508-R2(AMD)
Record Dates: First submitted 2025-08-06; First posted 2025-08-13 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: IBD - Inflammatory Bowel Disease; RA - Rheumatoid Arthritis
Keywords: pharmacokinetic-pharmacodynamic model; Model; IBD; Inflammatory Bowel Disease; Infliximab
MeSH Terms: conditions — Inflammatory Bowel Diseases; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with IBD: Patients who have active Crohn's disease with a score on the Crohn's disease activity index between 220 and 450 points. Or patient has active Ulcerative colitis defined by a total Mayo score between 6 and 12 points (part 2 only).
  Interventions: Drug: Subcutaneous infliximab CT-P13 Remsima®SC

INTERVENTIONS:
Drug: Subcutaneous infliximab CT-P13 Remsima®SC — Subcutaneous infliximab

SUMMARY:
A subcutaneous formulation of infliximab CT-P13 (Remsima, Celltrion) has been approved for clinical use in inflammatory bowel disease (IBD) and rheumatoid arthritis (RA) after demonstration of pharmacokinetic (PK) non-inferiority compared to intravenous CT-P13. The added value of the subcutaneous formulation of CT-P13 has been recognized by IBD physician expert, patients and nurses. However, further investigation is needed to select the right patients and timing for switching to the new subcutaneous formulation. Before investing resources into the design and execution of a prospective clinical trial to address these remaining clinical questions and concerns, an in silica simulation study using a population pharmacokinetic-pharmacodynamic (popPK-PD) model of CT-P13 would be highly informative. While popPK models of subcutaneous infliximab CT-P13 have been developed for both IBD and RA, a popPK-PD model is still awaited. The development of a popPK-PD model would allow us to bridge infliximab exposure and response, and address clinically relevant questions by focussing on therapeutic outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Crohns disease with a score on the Crohn's disease activity index between 220 and 450.
* Patients with active Ulcerative colitis as defined by a total Mayo score between 6 and 12 points (Part 2 only)

Exclusion Criteria:

* Patients who have previously received a biological agent for the treatment of CD and UC and/or a tumor necrosis factor-alpha (TNFa)-inhibitor for the treatment of other diseases.
* Patients who have allergies to any of the excipients of infliximab or any other murine and/or human proteins or patients with a hypersensitivity to immunoglobulin products.
* Patients who have a current or past history of infection with HIV, hepatitis B or C (carriers of hepatitis B and C are not permitted to enrol into the study, but past hepatitis B resolved can be enrolled).
* Patients who have acute infections requiring oral antibiotics within 2 weeks or parenteral injection of antibiotics within 4 weeks prior to the first administration of the study drug, other serious infection within 6 months prior to the first administration of the study drug or recurrent herpes zoster or other chronic or recurrent infection within 6 weeks prior to the first administration of the study drug.
* Patient who have an indeterminate result for interferon-y release assay (IGRA) or latent tuberculosis (TB) at Screening. For part 2, if IGRA result is indeterminate at the Screening, one retest will be possible during the screening. If the repeated IGRA result is negative, the patient can be included in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with inflammatory bowel disease
Sampling Method: Non-Probability Sample
Enrollment: 439 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Dose-exposure-response relationship of subcutaneous infliximab | At least 24 weeks
  To understand, describe, and predict the dose-exposure relationship of sibcutaneous infliximab in patients with inflammatory bowel diseased based on available data from previous clinical trials.

IPD SHARING:
Plan to Share IPD: Undecided
The decision that whether or not to share the IPD will depend of the modalities of the data transfer agreement.

REFERENCES:
- See also: Related Info — https://doi.org/10.1016/S0016-5085(23)03590-4
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/35390141/